CLINICAL TRIAL: NCT01456650
Title: Effect of the R230C Variant of the ATP-binding Cassette Transporter A1 (ABCA1) Gene on the Response to Treatment With Glibenclamide in Patients With Type 2 Diabetes Mellitus
Brief Title: R230C and C230C Variants of ABCA1 and Glyburide Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Carlos Aguilar, Vice Head of the Department of Endocrinology and Metabolism, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: INNSZ-ABCA1
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; ABCA1 alleles; Glyburide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glyburide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glyburide (Experimental): Patients in which the fasting glucose persisted above the treatment goal (fasting glucose <126 mg/dl) after a 4 week diet period will receive glyburide. The dose of the medication will be adjusted based on the results of fasting glucose values. At each visit patients will return the leftover tablets; counts of the tablets will be the method for measuring the adherence to treatment. The medical study participants who decided to doses of glibenclamide will not know the allele of ABCA1 gene under study.
  Interventions: Drug: Glyburide

INTERVENTIONS:
Drug: Glyburide — Patients in which the fasting glucose persisted above the treatment goal ( fasting plasma glucose above 126 mg/dl) will receive glyburide. The dose of the medication will be adjusted based on the result of blood glucose using the following table:
  Fasting glucose 126 to 140 mg/dl: 2.5 mg/day (half tablet in the morning) 141 to 180 mg/dl: 5 mg/day (a tablet in the morning) 181 220 mg/dl: 7.5 mg/day (a tablet in the morning and half tablet per night) 221 to 250 mg/dl: 10 mg/day (a tablet in the morning) and a tablet in the evening.

SUMMARY:
The objective of the study is to know if the R230C and C230C variants of the ATP-binding cassette transporter A1 (ABCA1) gene are associated with a smaller glucose lowering effect compared to the wild type allele (R230R) in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Specific objectives:

1. In patients with type 2 diabetes stratified by the existence of the risk alleles (R230C/C230C) or the wild variant (R230R) of ABC-A1, compare the changes resulting from the treatment with glibenclamide on following continuous variables:

   * Fasting glucose
   * Percentage reduction
   * Hemoglobin A1c,
   * Cholesterol, triglycerides, HDL cholesterol, LDL cholesterol
   * Weight
2. In patients with type 2 diabetes stratified by the existence of the risk alleles (R230C/C230C) or the wild variant (R230R) of ABC-A1, compare the changes resulting from the treatment with glibenclamide on following binomial variables:

   * Number of cases that reach fasting plasma glucose lower than 110 mg/dl
   * Number of cases that reach an HbA1c less than 7%

ELIGIBILITY:
Inclusion Criteria:

* Adults 20 to 79 years
* Body mass index >18 and 39.9 ≤
* Men or women
* Mexicans mestizos.
* Moderate hyperglycemia (126 to 250 mg/dl and HbA1c levels between 7 and 10%) despite being treated with a dietary program in combination or not with metformin (2 g/d).

Exclusion Criteria:

* Patients with chronic complications of diabetes: ischemic heart disease, stroke, proliferative retinopathy or blindness, albuminuria, chronic diarrhea, gastroparesis, non-traumatic amputation of lower limbs.
* Patients with any monogenic syndrome, obesity, diabetes or hypoalphalipoproteinemia
* Patients with acquired diseases that produce secondarily obesity or diabetes.
* Treatment with anorexigenics or accelerate weight loss at the time of the selection.
* Cardiovascular event in the 6 months prior to study entry.
* Steroids, chemotherapy, immunosuppressive or radiotherapy.
* Infections or concurrent acute diseases.
* Catabolic diseases such as cancer or AIDS
* Pregnancy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma fasting glucose | 20 weeks
  The effects of the alleles under study on the glucose lowering effect of glyburide will be assessed in 20 week study. Diet and exercise will be controlled per protocol

SECONDARY OUTCOMES:
HbA1c levels | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Aguilar-Salinas, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Aguilar-Salinas CA, Munoz-Hernandez LL, Cobos-Bonilla M, Ramirez-Marquez MR, Ordonez-Sanchez ML, Mehta R, Medina-Santillan R, Tusie-Luna MT. The R230C variant of the ATP binding cassette protein A1 (ABCA1) gene is associated with a decreased response to glyburide therapy in patients with type 2 diabetes mellitus. Metabolism. 2013 May;62(5):638-41. doi: 10.1016/j.metabol.2012.11.006. Epub 2012 Dec 27. PMID 23273975